CLINICAL TRIAL: NCT06606028
Title: Tumor-informed ctDNA Testing for Minimal Residual Disease Monitoring Following Curative-intent Treatment of Squamous Cell Carcinoma of the Head and Neck.
Brief Title: Tumor-Informed ctDNA Testing for MRD Following Treatment of Squamous Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Haystack Oncology, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 232010; NCI-2024-07739 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Squamous Cell Carcinoma of Head and Neck; Squamous Cell Carcinoma Head and Neck Cancer (HNSCC); Squamous Cell Carcinoma of Skin; Cutaneous Squamous Cell Carcinoma (CSCC)
Keywords: ctDNA
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Blood Specimen Collection; Histocompatibility Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue and blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Non-investigational Radiation therapy: Participants will have tumor tissue collected at screening and blood samples (approximately 20ml x 3) will be obtained during non-investigational, standard of care radiation and after care for up to 2 years.
  Interventions: Procedure: Blood Specimen Collection; Procedure: Tumor Tissue Collection; Other: Medical Record Review
- Cohort B: Non-investigational Surgery: Participants will have tumor tissue collected at screening and blood samples (approximately 20ml x 3) will be obtained during non-investigational, standard of care surgery and after care for up to 2 years.
  Interventions: Procedure: Blood Specimen Collection; Procedure: Tumor Tissue Collection; Other: Medical Record Review

INTERVENTIONS:
Procedure: Blood Specimen Collection — Approximately 20 mL of peripheral blood (10 mL per tube, x 3 Streck tubes) will be drawn at each time point
  Other Names: Blood Specimen; Biospecimen collection
Procedure: Tumor Tissue Collection — Formalin-fixed paraffin embedded tumor tissue samples (tissue blocks of 12 x 10 millimeter (mm) unstained slides) derived from biopsy or surgical resection will be collected at screening
  Other Names: Tissue Specimen; Biospecimen collection
Other: Medical Record Review — Medical records will be reviewed to collect standard of care p16 staining by immunohistochemistry and/or high-risk human papillomavirus (HPV) DNA or RNA testing that is performed as part of standard of care
  Other Names: Chart Review

SUMMARY:
This is a single-center, non-interventional, observational study that evaluates the correlation of circulating tumor DNA (ctDNA) testing to cancer relapse for participants with squamous cell carcinomas (HNC) of the head and neck mucosa and skin after curative-intent primary radiation or surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the rates of detectable ctDNA within two years of participants treated with curative-intent surgery or radiation-based treatment for HNC.

SECONDARY OBJECTIVES:

1. To describe the prevalence of detectable ctDNA at initial diagnosis in participants with HNC.
2. To describe the association of quantitative ctDNA levels with time-to-event outcomes (overall survival (OS), disease-free survival (DFS), and time to recurrence (TTR)).
3. To describe the association of quantitative ctDNA levels with follow-up imaging tumor volume.

OUTLINE:

Participants will have tissue samples collected at screening and blood samples collected for analysis before, during, and after non-investigational, standard of care treatment for cancer for up to 2 years

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically or cytologically confirmed squamous cell carcinoma of the head and neck mucosa and skin.
2. Participants must be age >=18 years.
3. Participants must be planning to receive curative-intent surgery or radiation-based treatment as part of standard of care treatment.
4. Participants must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Contraindication to phlebotomy for removal of 20 mL of peripheral blood each time point (up to 300 mL total over 15 time points).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with squamous cell carcinoma of the head and neck mucosa and skin.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence rate of ctDNA | Up to 2 years
  Cumulative incidence will be estimated by evaluating the cumulative incidence of positive ctDNA (non-zero) with death as a competing risk.

SECONDARY OUTCOMES:
Proportion of participants at diagnosis with a positive (non-zero) ctDNA result. | Up to 2 years
  The prevalence of detectable ctDNA at initial diagnosis in participants with locally-advanced head and neck cancer will be reported as the proportion of participants at diagnosis with a positive (non-zero) ctDNA result.
Association of association of quantitative ctDNA levels with overall survival (OS) | Up to 2 years
  The Spearman's correlation coefficient (rs) measures the strength and direction of association between two variables. The Spearman correlation coefficient, rs, can take values from +1 to -1 where a value of +1 indicates a perfect association, an rs of 0 indicates no association and an rs of -1 indicates a perfect negative association. The closer rs is to 0, the weaker the association. This correlation will be used to determine the association of quantitative ctDNA levels with overall survival (OS).
Association of association of quantitative ctDNA levels with disease-free survival (DFS) | Up to 2 years
  The Spearman's correlation coefficient (rs) measures the strength and direction of association between two variables. The Spearman correlation coefficient, rs, can take values from +1 to -1 where a value of +1 indicates a perfect association, an rs of 0 indicates no association and an rs of -1 indicates a perfect negative association. The closer rs is to 0, the weaker the association. This correlation will be used to determine the association of quantitative ctDNA levels with overall survival (OS).
Association of association of quantitative ctDNA levels with time to recurrence (TTR) | Up to 2 years
  The Pearson correlation coefficient (r) measures the strength and direction of association between two variables. The Pearson correlation coefficient (r) can take values from +1 to -1 where a value of +1 indicates a perfect association, a value of 0 indicates no association, and a value of -1 indicates a perfect negative association. The closer r is to 0, the weaker the association. This correlation will be used to determine the association of quantitative ctDNA levels with TTR.
Association of quantitative ctDNA levels with follow-up imaging tumor volume. | Up to 2 years
  The Pearson correlation coefficient (r) measures the strength and direction of association between two variables. The Pearson correlation coefficient (r) can take values from +1 to -1 where a value of +1 indicates a perfect association, a value of 0 indicates no association, and a value of -1 indicates a perfect negative association. The closer r is to 0, the weaker the association. This correlation will be used to determine the association of quantitative ctDNA levels with tumor volume.

CONTACTS AND LOCATIONS:
Overall Officials: Jason W Chan, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
De-identified laboratory data will be shared with industry collaborators on this study only